CLINICAL TRIAL: NCT06266858
Title: A Single-Center, Open-Label Study to Assess the Severity of Mitral Regurgitation With Multimodality Imaging
Brief Title: Multimodality Imaging Assessment of the Severity of Mitral Regurgitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Maohuan Lin, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SYSKY-2022-407-02
Record Dates: First submitted 2024-01-21; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Mitral Regurgitation
Keywords: mitral regurgitation; ultrasonic cardiography; cardiac magnetic resonance
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Fluid Therapy; Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- UCG in pre-anaesthetic group (Other): The fasting patients receive UCG in pre-anaesthetic.
  Interventions: Diagnostic Test: UCG; Other: fasting
- UCG in post-anaesthetic group (Other): The fasting patients receive UCG in post-anaesthetic.
  Interventions: Diagnostic Test: UCG; Other: fasting
- UCG in post-rehydration group (Other): The fasting patients in anaesthetised receive UCG in post-rehydration.
  Interventions: Other: rehydration; Diagnostic Test: UCG; Other: fasting
- cardiac magnetic resonance （CMR） group (Other): The non-fasting patients receive CMR in another time.
  Interventions: Diagnostic Test: CMR

INTERVENTIONS:
Other: rehydration — The fasting patients in anaesthetised receive saline rehydration to maintain central venous pressure of 6-8 cmH2O when undergoing UCG.
  Arms: UCG in post-rehydration group
Diagnostic Test: UCG — UCG is the most common imaging modality to assess the mitral regurgitation in clinical and also is the primary modality recommended by guidelines. At the beginning of the study, the fasting patients receive UCG in the different situation such as pre-anaesthetic, post-anaesthetic and post-rehydration.
  Arms: UCG in post-anaesthetic group; UCG in post-rehydration group; UCG in pre-anaesthetic group
Diagnostic Test: CMR — CMR may be more accurate than UCG in assessing MR severity. In another time, the patients receive CMR.
  Arms: cardiac magnetic resonance （CMR） group
Other: fasting — At the beginning of the study, the patients need to fast when receive UCG.
  Arms: UCG in post-anaesthetic group; UCG in post-rehydration group; UCG in pre-anaesthetic group

SUMMARY:
To investigate to assess the severity of mitral regurgitation by multimodality imaging.

DETAILED DESCRIPTION:
In the single-center and open-label study, the researcher will compare the changes of ultrasonic cardiography (UCG) parameters when patients in fasting, anaesthesia and rehydration firstly. The aims are to clarify the effect of fasting and anaesthesia on the assessment of mitral regurgitation (MR) severity and the corrective effect of intravenous rehydration. The researcher then will investigate the correlation and consistency of multimodality imaging in assessing the severity of mitral regurgitation. The aim is to acquire more accurate, objective and reproducible parameters, to provide new solution for the precise assessment of MR severity and to guide the selection of clinical treatment and timing.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years old
2. all-caused moderate or severe MR assessed by Trans-Thoracic Echocardiography (TTE) : 1) EROA ≥0.3cm^2; 2) RVol ≥45ml
3. The patient has signed an informed consent form.

Exclusion Criteria:

1. unstable angina, acute myocardial infarction and surgical history of coronary artery bypass grafting (CABG) and percutaneous coronary intervention (PCI) within 3 months before recruit
2. acute heart failure or acute worsening of chronic heart failure requiring vasoactive drug therapy
3. severe infections, septicaemia
4. severe hepatic insufficiency ( Child-Pugh class C)
5. severe renal insufficiency ( chronic kidney disease (CKD) stage 5: estimated glomerular filtration rate (eGFR) <15ml/min or dialysis)
6. hypotensive state, shock ( systolic blood pressure <90mmHg or mean arterial pressure <70mmHg with tissue hypoperfusion and urine output <30ml/h)
7. uncontrolled diseases of the haematological system: acute gastrointestinal bleeding, intracranial haemorrhage or haemorrhage from other organs, acute pulmonary embolism or deep vein thrombosis, congenital or acquired haemorrhagic disease such as haemophilia, anaphylactic purpura and acute leukaemia, severe abnormalities in haematological parameters such as platelet count <20*10^9/l and international normalized ratio (INR) >3
8. contraindication for Trans-Esophageal Echocardiography (TEE) such as oesophageal constriction, oesophageal tumour, oesophageal fistula, oesophageal varices, cervical vertebral instability
9. contraindication for CMR such as metal foreign matter in the body, claustrophobia
10. contraindication for intravenous anaesthesia such as allergy to anaesthetics
11. pregnancy or breastfeeding
12. The patient does not sign an informed consent form.
13. Due to other reasons the patient is not suitable for enrollment assessed by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
effective regurgitant orifice area (EROA) | 1 day during an examination
  EROA measured by multiple imaging methods when patient is in the different situation.
mitral regurgitant volume (RVol) | 1 day during an examination
  RVol measured by multiple imaging methods when patient is in the different
mitral regurgitant fraction (RF) | 1 day during an examination
  RF measured by multiple imaging methods when patient is in the different

CONTACTS AND LOCATIONS:
Overall Officials: Maohuan Lin, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China